CLINICAL TRIAL: NCT03842228
Title: A Phase 1b Biomarker-Driven Combination Trial of Copanlisib, Olaparib, and Durvalumab (MEDI4736) in Patients With Advanced Solid Tumors
Brief Title: Testing the Combination of the Anti-cancer Drugs Copanlisib, Olaparib, and MEDI4736 (Durvalumab) in Patients With Advanced Solid Tumors With Selected Mutations
Acronym: COD
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-00601; NCI-2019-00601 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI10217; 10217 (Other: University of Texas MD Anderson Cancer Center LAO); 10217 (Other: CTEP); UM1CA186688 (NIH)
Record Dates: First submitted 2019-02-07; First posted 2019-02-15 (Actual); Results first posted 2025-08-03 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Biopsy; Specimen Handling; copanlisib; durvalumab; Immunoglobulin G; Disulfides; Magnetic Resonance Spectroscopy; olaparib; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (copanlisib hydrochloride, olaparib, and durvalumab) (Experimental): See Detailed Description
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Copanlisib Hydrochloride; Biological: Durvalumab; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Drug: Olaparib; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Copanlisib Hydrochloride — Given IV
  Other Names: 5-Pyrimidinecarboxamide, 2-Amino-N-(2,3-dihydro-7-methoxy-8-(3-(4-morpholinyl)propoxy)imidazo(1,2-C)quinazolin-5-yl)-, Hydrochloride (1:2); Aliqopa; BAY 80-6946 Dihydrochloride; BAY-80-6946 Dihydrochloride; Copanlisib Dihydrochloride
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI 4736; MEDI-4736; MEDI4736
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
Procedure: X-Ray Imaging — Undergo x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase Ib trial seeks to identify the side effects and best dose of the combination of copanlisib and olaparib when given together with durvalumab. The trial will evaluate how well the drug combinations work in treating patients with advanced cancers who have solid tumors that have spread from where they first started (primary site) to other places in the body (metastatic) or cannot be removed by surgery (unresectable). Copanlisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. PARPs are proteins that help repair DNA mutations. PARP inhibitors, such as olaparib, can keep PARP from working, so tumor cells can't repair themselves and may stop growing. Immunotherapy with monoclonal antibodies, such as durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. The treatment combinations of copanlisib and olaparib or copanlisib, olaparib, and durvalumab may work better in treating patients with solid tumors compared to usual treatments such as surgery, radiation, or other chemotherapy drugs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and establish the recommended phase 2 dose (RP2D) of the doublet combination of copanlisib and olaparib and of the triplet combination of copanlisib, olaparib and MEDI4736 (durvalumab) in patients with molecularly-selected solid tumors.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity of the doublet combination of copanlisib and olaparib, and of the triplet combination of copanlisib, olaparib and MEDI4736 (durvalumab) in patients with molecularly-selected advanced solid tumors, as measured by objective response rate (ORR) (complete response [CR] + partial response [PR]). Although the clinical benefit of the doublet and triplet combination of these drugs has not yet been established, the intent of offering this treatment is to provide a possible therapeutic benefit, and thus the patient will be carefully monitored for tumor response and symptom relief in addition to safety and tolerability.

II. To assess overall duration of response (DoR), progression free survival (PFS) and overall survival (OS).

III. To assess the pharmacokinetic (PK) profiles of these combinations, and explore exposure-response relationships.

IV. To correlate molecular alterations with OR (CR+PR).

OUTLINE: This is a dose-escalation and expansion study of the doublet combination of copanlisib and olaparib or the triplet combination of copanlisib, olaparib, durvalumab.

In the dose escalation phase of the study, patients treated with the doublet combination will receive copanlisib hydrochloride intravenously (IV) over 1 hour on days 1 and 15 or days 1, 8, and 15 depending on dose level and olaparib orally (PO) twice daily (BID) on days 1-28 of each cycle. Patients treated with the triplet combination will also receive copanlisib hydrochloride and olaparib, in addition to also receiving durvalumab beginning in cycle 2. Beginning in cycle 2, patients treated with the triplet combination will receive durvalumab IV over 1 hour on day 1 of each cycle. In the dose expansion phase of the study, patients will be treated with the best study drug dose identified in the dose escalation phase of the study.

For all patients treated with the doublet and triplet combinations, the cycles will repeat every 28 days for 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples at baseline within 7 days of cycle 1 day 1 (C1D1), days 8 and 15 of cycle 1 and day 15 of subsequent cycles, at time of restaging, and end of treatment/progression. Patients undergo x-ray, computed tomography (CT), and magnetic resonance imaging (MRI) at the end of cycle 2 and then every 8 weeks. Patients also undergo an echocardiography (ECHO) during pre-study within 28 days of C1D1 and tumor biopsy at baseline within 7 days of C1D1 and day 15 of cycle 1 or 2, and may undergo an optional biopsy at end of treatment/progression.

After completion of study treatment, all patients are followed up at 30 days and then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* ELIGIBILITY CRITERIA FOR ENROLLMENT INTO STEPS 1, 2, AND 3
* Patients must have germline or somatic mutations in DDR genes: BARD1, BRCA1, BRCA2, BRIP1, FANCA, NBN, PALB2, RAD51, RAD51B, RAD51C, RAD51D; or actionable mutations in the PTEN gene, or hotspot mutations in the PIK3CA gene (E542, E545 or H1047 are accepted). Local testing in Clinical Laboratory Improvement Act (CLIA)-certified laboratory will be accepted. Only mutations that have been recognized as actionable by the MD Anderson Precision Oncology Decision Support (PODS) team will be accepted
* Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Patients must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Patients must be >= 3 weeks beyond treatment with any chemotherapy or >= 4 weeks beyond treatment with other investigational therapy to include hormonal, biological, or targeted agents; or at least 5 half-lives from hormonal, biological, or targeted agents, whichever is shorter at the time of treatment initiation
* Age >= 18 years. Because no dosing or adverse event (AE) data are currently available on the use of copanlisib in combination with olaparib +/- durvalumab (MEDI4736) in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Patients with a mutation within both the DDR and PTEN/PIK3CA pathways will be assessed by the genomics Precision Oncology Decision Support group at MD Anderson, and the patient will be allocated to the PI3K or DDR expansion group deemed to be the main driver. If the actionability between the groups is deemed to be equivocal, then the patient will be allocated to the expansion cohort with fewer patients
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 1 (Karnofsky >= 60%)
* Hemoglobin >= 10 g/dL with no blood transfusion in the past 28 days
* Leukocytes >= 3,000/mcL
* Lipase =< 1.5 x upper limit of normal (ULN)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 140,000/mcL
* Total bilirubin =< 1.5 x institutional ULN
* Serum bilirubin =< 1.5 x institutional ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN, unless liver metastases are present in which case they must be =< 5 x ULN
* Activated partial thrombin time =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as prothrombin time (PT) or partial thromboplastin time (PTT) is within the therapeutic range of intended use of anticoagulants
* International normalized ratio =< 1.5 x ULN
* Glomerular filtration rate (GFR) >= 51 mL/min, based on a 24-hour urine test for creatinine clearance or estimated using the Cockcroft-Gault equation
* Left ventricular ejection fraction (LVEF) >= 50%
* Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that their medication dose and international normalized ratio (INR)/PTT is stable
* Prophylactic antiemetics may be administered according to standard practice. The routine use of standard antiemetics, including 5-hydroxytryptamine type 3 (5-HT3) blockers, such as granisetron, ondansetron, or an equivalent agent, is allowed as needed. The use of corticosteroids as antiemetics prior to copanlisib administration will not be allowed
* Postmenopausal or evidence of non-childbearing status, a negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1. Postmenopausal is defined as:

  * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
  * Luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the postmenopausal range for women under 50
  * Radiation-induced oophorectomy with last menses > 1 year ago
  * Chemotherapy-induced menopause with > 1 year interval since last menses
  * Surgical sterilization (bilateral oophorectomy or hysterectomy)
* Women of child-bearing potential MUST have a negative serum or urine human chorionic gonadotropin (HCG) test unless prior tubal ligation (>= 1 year before screening), total hysterectomy or menopause (defined as 12 consecutive months of amenorrhea). Patients should not become pregnant or breastfeed while on this study
* Patients and their partners, if sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in combination throughout the period of taking study treatment and for 6 months after last dose of study drug(s) to prevent pregnancy in the study patient or partner. Male patients should avoid donating sperm for 3 months following the last dose of olaparib
* Human immunodeficiency virus (HIV)-infected (HIV 1/2 antibody-positive; HIV testing pre-study not required) patients may participate IF they meet all the following eligibility requirements:

  * They must be on an anti-retroviral regimen with evidence of at least two undetectable viral loads within the past 6 months on this same regimen; the most recent undetectable viral load must be within the past 12 weeks
  * They must have a CD4 count >= 250 cells/mcL over the past 6 months on this same anti-retroviral regimen and must not have had a CD4 count < 200 cells/ mcL over the past 2 years, unless it was deemed related to the cancer and/or chemotherapy-induced bone marrow suppression

    * For patients who have received chemotherapy in the past 6 months, a CD4 count < 250 cells/mcL during chemotherapy is permitted as long as viral loads were undetectable during this same chemotherapy
  * They must have an undetectable viral load and a CD4 count >= 250 cells/mcL within 7 days of enrollment
  * They must not be currently receiving prophylactic therapy for an opportunistic infection and must not have had an opportunistic infection within the past 6 months
* Ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) must have a legally authorized representative or caregiver who gives such consent
* Patient is willing and able to comply with the protocol for the duration of the study, including undergoing treatment and scheduled visits and examinations
* Patients with a tumor that is readily accessible for biopsy
* ELIGIBILITY CRITERIA FOR ENROLLMENT INTO STEP 2 AND 3 ONLY
* Body weight > 30 kg
* Life expectancy >= 16 weeks

Exclusion Criteria:

* EXCLUSION CRITERIA FOR STEPS 1, 2, AND 3
* Persistent toxicities (> Common Terminology Criteria for Adverse Events [CTCAE] grade 2) caused by previous cancer therapy, excluding alopecia
* Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery
* Patients who are receiving any other investigational agents
* Other malignancy unless curatively treated with no evidence of disease for >= 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), or stage 1, grade 1 endometrial carcinoma. A patient with a history of localized triple negative breast cancer may be eligible, provided the patient completed the adjuvant chemotherapy > 3 years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients with myelodysplastic syndrome/acute myeloid leukemia (MDS/AML) or with bone marrow findings consistent with MDS/AML
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib, copanlisib, PI3K inhibitors or MEDI4736 (durvalumab) or any of the excipients of any study products
* Concomitant use of strong CYP3A inhibitors and inducers

  * Olaparib: concomitant use of known strong CYP3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g., ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period for strong or moderate CYP3A inhibitors prior to starting olaparib is 2 weeks
  * Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
  * Concomitant use of known strong CYP3A inducers (e.g., phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g., bosentan, efavirenz, modafinil). The required washout period for strong or moderate CYP3A inducers prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents
  * Copanlisib: copanlisib is primarily metabolized by CYP3A4. Therefore, the concomitant use of strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir and saquinavir), and strong inducers of CYP3A4 (e.g. rifampin, phenytoin, carbamazepine, phenobarbital, St. John's Wort) are not permitted from 14 days prior to enrollment until the end of the study
  * Other medications that are prohibited while on copanlisib treatment:

    * Herbal medications/preparations (except for vitamins)
    * Anti-arrhythmic therapy other than beta blockers or digoxin
  * Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference for a list of drugs to avoid or minimize use of. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan, symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Resting electrocardiogram (ECG) indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QT corrected by the Fridericia formula [QTcF] prolongation of > 500 msec, electrolyte disturbances), or patients with congenital long QT syndrome
* Women who are breast feeding or pregnant are excluded from this study because olaparib is a poly (adenosine diphosphate-ribose) polymerase (PARP) inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with olaparib, breastfeeding should be discontinued if the mother is treated with olaparib and copanlisib +/- MEDI4736 (durvalumab)
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Packed red blood cell or platelet transfusion in the last 28 days prior to study entry
* Whole blood transfusions in the last 120 days prior to study entry. Whole blood transfusions performed within 120 days of study entry may interfere with blood samples taken for exploratory analysis
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. However, systemic corticosteroids may be indicated after starting the study drugs to treat immune-related adverse reactions. Inhaled or topical steroids and adrenal replacement doses =< 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Patients with non-healing wound, ulcer, or bone fracture
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before the start of study medication
* Patients with active, clinically serious infections > grade 2 (CTCAE version[v] 5.0). Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis [TB] testing in line with local practice), hepatitis B (known positive hepatitis B virus [HBV] surface antigen [HBsAg] result), or hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA). HBV/HCV screening is required 28 days prior to starting the study drug using a routine hepatitis virus lab panel
* Active infection requiring IV antibiotics or other uncontrolled intercurrent illness requiring hospitalization
* Patients unable to swallow orally administered medication and any medical condition or diagnosis that would likely impair absorption of an orally administered drug (e.g. gastrectomy, ileal bypass, chronic diarrhea, gastroparesis)
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* New York Heart Association class III or IV heart disease
* History or concurrent interstitial lung disease of any severity and/or severely impaired lung function (as judged by the investigator)
* Uncontrolled arterial hypertension despite optimal medical management (per investigator's opinion)
* Patients with uncontrolled type I or II diabetes mellitus, defined as fasting blood glucose ˃ 160 mg/dL and glycosylated hemoglobin (HbA1c) ˃ 8%, are ineligible
* EXCLUSION STEPS 2 AND 3 ONLY
* Patients who have not recovered from grade >= 2 adverse events due to prior anti-cancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

  * Patients with grade >= 2 neuropathy will be evaluated on a case-by-case basis after consultation with the study physician
* Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of investigational product (IP). Note: local surgery of isolated lesions for palliative intent is acceptable
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP
* Patients with unstable angina pectoris
* Patients who have received prior anti-PD-1, anti PD-L1 or anti CTLA-4:

  * Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy. All adverse events (AEs) while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study
  * Must not have experienced a grade >= 3 immune-related AE or an immune-related neurologic or ocular AE of any grade while receiving prior immunotherapy. Note: Patients with an endocrine AE of grade =< 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic
  * Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day
* Live vaccination, including virus vaccination and yellow fever vaccination, within 6 months before start of study treatment
* Cytomegalovirus (CMV) infection. Patients who are known to be CMV polymerase chain reaction (PCR) positive at baseline will not be eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2026-09-24 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A Yap, Principal Investigator — University of Texas MD Anderson Cancer Center LAO
Locations (17):
- United States (17):
  - Keck Medicine of USC Buena Park, Buena Park, California
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Texas at Austin, Austin, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase Ib multicenter study led by MD Anderson Cancer Center. Participants were eligible if they had (1) advanced solid tumors for which curative measures did not exist or were no longer effective and (2) an actionable mutation in DNA Damage Response (DDR) genes (BARD1, BRCA1,BRCA2, BRIP1, FANCA, NBN, PALB2, RAD51, RAD51B, RAD51C, RAD51D), PTEN, or PIK3CA hotspots (E542, E545, or H1047).
Pre-assignment Details: Patients were enrolled into the following cohorts: Step 1 (Copanlisib and Olaparib dose escalation), Step 2 (Copanlisib, Olaparib, and Durvalumab dose escalation), or Step 3 (Copanlisib and Olaparib dose expansion). Patients enrolled in Step 3 were enrolled in the following dose expansion sub-cohorts: (1) those with germline or somatic DDR mutations (the DDR arm) or (2) those with PIK3CA or PTEN mutations (PIK3CA/PTEN arm). Thirty-nine patients were treated in Steps 1 - 3.
Groups:
- Step 1 Dose Level 1: Step 1 DL1: Copanlisib 45 mg IV (days 1, 8, 15) + Olaparib 200 mg PO BID; 28-day cycle
- Step 1 Dose Level 2: Step 1 DL2: Copanlisib 45 mg IV (days 1, 8, 15) + Olaparib 300 mg PO BID; 28-day cycle
- Step 1 Dose Level 3: Step 1 DL3: Copanlisib 60 mg IV (days 1, 8, 15) + Olaparib 300 mg PO BID; 28-day cycle
- Step 1 Dose Level 3A: Step 1 DL3A: Copanlisib 60 mg IV (days 1 and15) + Olaparib 300 mg PO BID; 28-day cycle
- Step 2 Dose Level 1: Step 2 DL1:
  Copanlisib 60 mg IV (days 1 and15) + Olaparib 300 mg PO BID + Durvalumab 1500 mg IV on day 1 starting at C2D1 ; 28-day cycle"
- Step 3 DDR Arm; Step 3 PIK3CA/PTEN Arm: Step 3 DL3A: Copanlisib 60 mg IV (days 1 and15) + Olaparib 300 mg PO BID; 28-day cycle
Period: Overall Study
Arm/Group | Step 1 Dose Level 1 | Step 1 Dose Level 2 | Step 1 Dose Level 3 | Step 1 Dose Level 3A | Step 2 Dose Level 1 | Step 3 DDR Arm | Step 3 PIK3CA/PTEN Arm
Started | 9 | 3 | 10 | 6 | 4 | 2 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 9 | 3 | 10 | 6 | 4 | 2 | 5
Not completed — Adverse Event | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1 | 0 | 0 | 2
Not completed — Progression | 8 | 1 | 7 | 5 | 4 | 2 | 3

BASELINE CHARACTERISTICS:
Population: All 39 patient treated on-study in Steps 1-3
Groups:
- Total: Total of all reporting groups
Arm/Group | Step 1 Dose Level 1 | Step 1 Dose Level 2 | Step 1 Dose Level 3 | Step 1 Dose Level 3A | Step 2 Dose Level 1 | Step 3 DDR Arm | Step 3 PIK3CA/PTEN Arm | Total
Number analyzed (Participants) | 9 | 3 | 10 | 6 | 4 | 2 | 5 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 1 | 8 | 3 | 4 | 2 | 3 | 27
  >=65 years | 3 | 2 | 2 | 3 | 0 | 0 | 2 | 12
Age, Continuous [Median (Full Range); unit: years] | 63 [29 to 70] | 67 [52 to 76] | 59 [46 to 67] | 63.5 [28 to 74] | 51 [35 to 60] | 44.5 [37 to 52] | 64 [58 to 83] | 60 [28 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7 | 6 | 3 | 2 | 2 | 27
  Male | 3 | 2 | 3 | 0 | 1 | 0 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 9 | 3 | 8 | 5 | 4 | 2 | 4 | 35
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 3
  White | 9 | 3 | 8 | 4 | 4 | 1 | 5 | 34
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 3 | 10 | 6 | 4 | 2 | 5 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicities (DLT) as a Measure of Safety Profile to Determine Recommended Phase 2 Dose (RP2D)
Description: A DLT was evaluated according to the NCI CTCAE 5.0. An AE was defined as DLT if it met any of the following events: any grade 5 toxicity; any grade 2 toxicity that require permanent discontinuation of durvalumab or combination therapies within the first 4 weeks; grade 4 neutropenia; febrile neutropenia; neutropenic infection; grade ≥ 3 thrombocytopenia with bleeding; grade 4 thrombocytopenia; Grade 4 anemia; non-hematological grade ≥ 4 toxicities; confirmation of QTc prolongation; grade ≥3 AE hyperglycemia or hypertension lasting < 7 days; grade 3 skin rash despite optimal medical intervention; grade 3 diarrhea despite optimal medical intervention; any toxicity greater than baseline & clinically significant or unacceptable & disrupts dosing for more than 14 days; any event, including significant dose reductions or omissions as judged by safety review committee; & any toxicity in any course of treatment that in the opinion of the investigators and medical monitors is dose-limiting.
Time Frame: The DLT monitoring time frame was Cycle 1 through Cycle 2 Day 1 for the doublet combination (SIL1, SIL2, SIL3, and SIL3A) , and Cycle 1 through Cycle 3 Day 1 for the triplet combination (S2L1)
Population: To be evaluable for DLT, patients must receive at least 75% of Olaparib doses and have no missed Copanlisib doses. In Step 1 dose level 3, Step 1 dose level 3A, Step 2 dose level 1, and Step 3 PIK3CA/PTEN arm, 8 patients were not evaluable for DLT because they did not receive sufficient drug in Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Step 1 Dose Level 1 | Step 1 Dose Level 2 | Step 1 Dose Level 3 | Step 1 Dose Level 3A | Step 2 Dose Level 1 | Step 3 DDR Arm | Step 3 PIK3CA/PTEN Arm
Number analyzed (Participants) | 9 | 3 | 10 | 6 | 4 | 2 | 5
Participants
  DLT | 1 | 0 | 2 | 0 | 0 | 0 | 0
  No DLT | 8 | 3 | 4 | 5 | 3 | 2 | 3
  Not evaluable for DLT | 0 | 0 | 4 | 1 | 1 | 0 | 2

2. Secondary Outcome: Objective Response Rate (ORR = Complete Response [CR] + Partial [PR])
Description: Anti-tumor activity of the combination of copanlisib and olaparib, and of the triplet combination of copanlisib, olaparib, and durvalumab will be measured by ORR. Will estimate ORR with 95% confidence intervals.
Time Frame: Up to 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Duration of Response
Description: Will use the Kaplan-Meier method to estimate this distribution.
Time Frame: From time measurement criteria are met for CR or PR until the first date that recurrent or progressive disease is objectively documented, assessed up to 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Progression-free Survival
Description: Will use the Kaplan-Meier method to estimate this distribution.
Time Frame: From start of treatment to time of progression or death, whichever occurs first, assessed up to 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival
Description: Will use the Kaplan-Meier method to estimate this distribution.
Time Frame: Up to 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Pharmacokinetics of Copanlisib and Olaparib (Doublet Combination); Step 1 Cohorts
Description: Assessment of pharmacokinetic profiles of copanlisib and olaparib at various treatment timepoints.
Time Frame: Step 1: C1D8- baseline; 30 and 55 mins post start copanlisib(copa),1 hour (h), 3h, 5h, 7h, and 23h after end of copa; C1D15: baseline, 30 min, 55min post start copa infusion. Step 1 DL3A: only C1D15 timepoints.
Reporting Status: Not Posted

7. Secondary Outcome: Pharmacokinetics Off Copanlisib, Olaparib, and Durvalumab (Triplet Combination); Step 2 Cohorts
Description: Assessment of pharmacokinetic profiles of copanlisib, olaparib, and durvalumab at various treatment timepoints.
Time Frame: Cycle 1, day 15: baseline (predose), 30 min, 55 min post start copanlisib infusion, and 1 h, 3h, 5h, 7h, and 23h post end of copanlisib infusion, Day 1 on cycles 2-5: baseline (predose) and 50 min post start of durvalumab infusion
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Approximately four years and eight months, from the time the first patient signed the informed consent, throughout the treatment period, and up to 90 days after the administration of the last dose of study drug.
Description: Incidence and causality of all adverse events (AE) of all grades and attribution for all patients treated on-study, and were graded based on the Common Terminology Criteria for Adverse Events (CTCAE) version 5. All advserse events were captured from the time of signing consent through 90 days after the administration of the last dose of study drug. Only the highest graded AE per patient was evaluated per AE event term listed below.
Arm/Group | Step 1 Dose Level 1 | Step 1 Dose Level 2 | Step 1 Dose Level 3 | Step 1 Dose Level 3A | Step 2 Dose Level 1 | Step 3 DDR Arm | Step 3 PIK3CA/PTEN Arm
All-Cause Mortality (participants affected / at risk) | 9/9 | 1/3 | 8/10 | 2/6 | 2/4 | 0/2 | 2/5
Serious Adverse Events (participants affected / at risk) | 5/9 | 1/3 | 5/10 | 5/6 | 3/4 | 2/2 | 5/5
Other Adverse Events (participants affected / at risk) | 9/9 | 3/3 | 10/10 | 6/6 | 4/4 | 2/2 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1 Dose Level 1 (N=9) | Step 1 Dose Level 2 (N=3) | Step 1 Dose Level 3 (N=10) | Step 1 Dose Level 3A (N=6) | Step 2 Dose Level 1 (N=4) | Step 3 DDR Arm (N=2) | Step 3 PIK3CA/PTEN Arm (N=5)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
ALT increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
AST increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Esophageal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Fever (General disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1 Dose Level 1 (N=9) | Step 1 Dose Level 2 (N=3) | Step 1 Dose Level 3 (N=10) | Step 1 Dose Level 3A (N=6) | Step 2 Dose Level 1 (N=4) | Step 3 DDR Arm (N=2) | Step 3 PIK3CA/PTEN Arm (N=5)
Anemia (Blood and lymphatic system disorders) | 2 | 3 | 3 | 2 | 2 | 1 | 3
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 1 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Allergic reaction (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
ALT increased (Investigations) | 2 | 0 | 3 | 0 | 2 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 4 | 3 | 1 | 1
Anxiety (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
AST increased (Investigations) | 2 | 0 | 3 | 0 | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 0
Bacteremia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bloating (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Blood bukurubin increased (Investigations) | 0 | 0 | 3 | 0 | 0 | 0 | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 3 | 2 | 5 | 1 | 1 | 0 | 1
Blood/lymph - Other - Mild Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blurred vision (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac troponin I increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Confusion (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 2 | 1 | 4 | 3 | 1 | 1
Corneal ulcer (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 3 | 0 | 1
Creatinine increased (Investigations) | 3 | 2 | 3 | 1 | 2 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 1 | 5 | 5 | 1 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 2
Dry Eye (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Dysesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 2 | 2 | 1 | 0 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 5 | 2 | 1 | 2
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Ear and labyrinth - other - Phonophobia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Edema limbs (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Elevated LDH (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Esophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye disorders - Other, specify - ocular erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, specify - stye (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye disorders - Other, specify - Subjunctival Hemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, specify - Swollen (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid function disorder (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Fatigue (General disorders) | 3 | 0 | 2 | 4 | 1 | 2 | 4
Fever (General disorders) | 2 | 0 | 4 | 1 | 2 | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Flu like symptoms (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Fracture (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Generalized edema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
GI disorders - Other, specify - Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
GI disorders - Other, specify - Stomach Bug (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
GI disorders - Other, specify - Swollen Tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 2 | 1 | 0 | 0 | 1
Hemmorrhoids (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 4 | 3 | 1 | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 3 | 0 | 2 | 5 | 2 | 1 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 0 | 3 | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1
Hypoatremia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 1 | 1 | 1 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 3
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypothyroidism (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Ilean ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infections & infestations - Other - Kidney Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infections & infestations - Other - Picc Line Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infections & infestations - Other - Sars-Cov-2 Virus (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infections & infestations - Other - Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infections & infestations - Other - Tumor Necrosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (General disorders) | 1 | 1 | 1 | 1 | 2 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metabolism and nutrition - Other - Iron Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 4 | 2 | 4 | 2 | 1 | 0 | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 2 | 5 | 5 | 4 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Night blindness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 1 | 3 | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Phantom pain (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photophobia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 2 | 2 | 1 | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2
portal vein thrombosis (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Pruitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 2 | 4 | 3 | 2 | 1 | 3
Rectal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal & urinary disorders - Other - Incomplete Voiding (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Reproductive and breast - Other - Uterine Fibroid (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Resp, thoracic & mediast - Other - Dry Mucous Membrane To Nose And Mouth (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Serum amylase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 4 | 2 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 0 | 0
Skin & subcutaneous tissue -Other - Buttock Skin Irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin & subcutaneous tissue -Other - Hand Blisters (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin & subcutaneous tissue -Other - Skin Changes, Pathches (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin & subcutaneous tissue -Other - Tick Bite (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Skin ulceration (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Superficial thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Surgical and medical - Other - Blepharoplasty (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Surgical and medical - Other - Bronchoscopy (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Surgical and medical - Other - Gastrointestinal Endoscopy (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Surgical and medical - Other - Insertion Of 4 Fr Double (Lumen Left Brachial Picc) (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Surgical&medical-Other-Insertion Of Tunneled Centrally Inserted Central Venous Catheter w/SQ port (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Surgical and medical - Other - Ir Transjugular Liver Biopsy (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Surgical and medical - Other - Lumbar Puncture (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Surgical and medical - Other - Nephrostomy Exchange (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Surgical and medical - Other - Nephrostomy Tube Placement (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Surgical and medical - Other - Nephrostomy Unilateral Placement (Hepatic Arterial Embolization) (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Surgical and medical - Other - Paracentesis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Surgical and medical - Other - Picc Insertion (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Surgical and medical - Other - Port-A-Cath Placement (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Surgical and medical - Other - Punch Biopsy Of Left Hand (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Surgical and medical - Other - Stent (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Surgical and medical - Other - Suture Removal Of Left Hand (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Surgical and medical - Other - Tooth Extraction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 2
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal discharge (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 0 | 1 | 0
Weight Loss (Investigations) | 0 | 1 | 0 | 3 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell decreasing (Investigations) | 1 | 2 | 1 | 1 | 1 | 0 | 0
Watering eyes (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT03842228/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT03842228/ICF_001.pdf